CLINICAL TRIAL: NCT03529110
Title: A Phase 3, Multicenter, Randomized, Open-Label, Active-Controlled Study of DS-8201a (Trastuzumab Deruxtecan), an Anti-HER2 Antibody Drug Conjugate (ADC), Versus Ado Trastuzumab Emtansine (T-DM1) for HER2-Positive, Unresectable and/or Metastatic Breast Cancer Subjects Previously Treated With Trastuzumab and Taxane
Brief Title: DS-8201a Versus T-DM1 for Human Epidermal Growth Factor Receptor 2 (HER2)-Positive, Unresectable and/or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane [DESTINY-Breast03]
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-U302; 2018-000222-61 (EudraCT Number); jRCT2080223919 (Registry Identifier: JAPIC CTI); DESTINY-B03 (Other: Daiichi Sankyo and AstraZeneca); CTR20190378 (Registry Identifier: CDE); 2024-511204-16-00 (EU CTIS Number)
Record Dates: First submitted 2018-04-13; First posted 2018-05-18 (Actual); Results first posted 2022-04-29 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Metastatic breast cancer; DS-8201a; DESTINY - Breast 03
MeSH Terms: conditions — Breast Neoplasms | interventions — trastuzumab deruxtecan; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Trastuzumab deruxtecan (T-DXd) (Experimental): Participants with HER2-positive, unresectable and/or metastatic breast cancer participants previously treated with trastuzumab and taxane who received T-DXd as a sterile intravenous (IV) solution at a dose of 5.4 mg/kg every 3 weeks (Q3W).
  Interventions: Drug: Trastuzumab deruxtecan (T-DXd)
- Ado-trastuzumab emtansine (T-DM1) (Active Comparator): Participants with HER2-positive, unresectable and/or metastatic breast cancer participants previously treated with trastuzumab and taxane who received T-DM1 in accordance with the approved label.
  Interventions: Drug: Ado-trastuzumab emtansine (T-DM1)

INTERVENTIONS:
Drug: Trastuzumab deruxtecan (T-DXd) — T-DXd is sterile lyophilized powder reconstituted into a sterile aqueous solution (100 mg/5 mL) to be administered intravenously.
  Other Names: DS-8201a
  Arms: Trastuzumab deruxtecan (T-DXd)
Drug: Ado-trastuzumab emtansine (T-DM1) — The treatment will be in accordance with the approved label.
  Other Names: T-DM1
  Arms: Ado-trastuzumab emtansine (T-DM1)

SUMMARY:
This study is designed to compare the anti-tumor activity as well as the safety and efficacy of DS-8201a versus T-DM1 in HER2-positive, unresectable and/or metastatic breast cancer subjects previously treated with trastuzumab and taxane.

ELIGIBILITY:
Inclusion Criteria:

1. Must be competent and able to comprehend, sign, and date an Institutional Review Board (IRB) or Ethics Committee (EC) approved ICF before performance of any study-specific procedures or tests.
2. Adults ≥18 y old. (Please follow local regulatory requirements if the legal age of consent for study participation is >18 y old.)
3. Pathologically documented breast cancer that:

   1. is unresectable or metastatic.
   2. has confirmed HER2-positive expression as determined according to American Society of Clinical Oncology - College of American Pathologists guidelines evaluated at a central laboratory.23
   3. was previously treated with trastuzumab and taxane in the advanced/ metastatic setting or progressed within 6 mo after neoadjuvant or adjuvant treatment involving a regimen including trastuzumab and taxane.
4. Documented radiologic progression (during or after most recent treatment or within 6 mo after completing adjuvant therapy).
5. Subjects must be HER2-positive as confirmed by central laboratory assessment of most recent tumor tissue sample available. If archived tissue is not available, a fresh biopsy is required.
6. Presence of at least 1 measurable lesion per modified Response Evaluation Criteria in Solid Tumors (mRECIST) version 1.1

Exclusion Criteria:

1. Prior treatment with an anti-HER2 ADC (such as T-DM1) in the metastatic setting. Prior treatment in the adjuvant/neoadjuvant setting would be allowed if progression of disease did not occur within 12 mo of end of adjuvant therapy.
2. Uncontrolled or significant cardiovascular disease, including any of the following:

   1. History of myocardial infarction within 6 mo before randomization;
   2. History of symptomatic congestive heart failure (New York Heart Association Class II to IV);
   3. Troponin levels consistent with myocardial infarction as defined according to the manufacturer within 28 d prior to randomization;
   4. Corrected QT interval (QTc) prolongation to > 470 ms (females) or >450 ms (male) based on average of Screening triplicate 12-lead ECG;
   5. LVEF < 50% within 28 d prior to randomization
3. Has a history of (noninfectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
4. Spinal cord compression or clinically active central nervous system (CNS) metastases, defined as untreated or symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.

   * Subjects with clinically inactive brain metastases may be included in the study.
   * Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 wk must have elapsed between the end of whole brain radiotherapy and study enrollment.
5. Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients in the drug product.
6. History of severe hypersensitivity reactions to other mAbs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2026-07-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Global Team Leader, Study Director — Daiichi Sankyo
Locations (164):
- United States (28):
  - UCLA Hematology Oncology, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Innovative Clinical Research Institute, Whittier, California
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - Florida Cancer Specialists-Broadway, Fort Myers, Florida
  - Florida Cancer Specialists NORTH, St. Petersburg, Florida
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - Loyola University Health System, Maywood, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - North Shore Hematology Oncology Associates, PC, East Setauket, New York
  - University of Rochester, Rochester, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Seidman Cancer Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Dayton Physicians, LLC, Kettering, Ohio
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - Tennessee Oncology- St Thomas Location, Nashville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital / Houston Methodist Cancer Center, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Millennium Oncology, Houston, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - MultiCare Health System Institute for Research and Innovation, Auburn, Washington
- Australia (6):
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Peninsula and South Eastern Haematology & Oncology Group, Frankston, Victoria
  - Peter MacCallum Cancer, Melbourne, Victoria
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- Belgium (6):
  - Institut Jules-Bordet, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Sint-Lucas - Campus Sint-Lucas, Ghent
  - Universitaire Ziekenhuizen Leuven, Leuven
  - CHU UCL Namur site de Sainte Elisabeth, Namur
- Brazil (8):
  - NOB - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul
  - Catarina Pesquisa Clinica, Itajaí, Santa Catarina
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André, São Paulo
  - ICESP - Instituto do Cancer do Estado de São Paulo Octavio Frias de Oliveira, São Paulo, São Paulo
  - Clínica de Pesquisas e Centro de Estudos em Oncologia Ginecológica e Mamária Ltda., São Paulo, São Paulo
  - Instituto Americas, Rio de Janeiro
  - A. C. Camargo Cancer Center, São Paulo
- Canada (3):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - St. Mary's Hospital, Montreal, Quebec
- China (12):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University, Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital Xiasha Branch, Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- France (22):
  - Centre Paul Strauss, Strasbourg, Bas Rhin
  - Hôpital Nord - CHU Marseille, Marseille, Bouches-du-Rhone
  - Centre François Baclesse, Caen, Calvados
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans, Cedex 02, Sarthe
  - CARIO - Centre Armoricain de Radiothérapie, Imagerie médicale et Oncologie, Plérin, Cotes d'Armor
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - CHRU Jean Minjoz, Besançon, Doubs
  - Institut Bergonié, Bordeaux, Gironde
  - Centre René Huguenin, Saint-Cloud, Hauts De Seine
  - ICM Val d'Aurelle, Montpellier, Herault
  - CRLCC Eugene Marquis, Rennes, Ille Et Vilaine
  - ICO - Site René Gauducheau, Saint-Herblain, Loire Atlantique
  - ICO - Site Paul Papin, Angers, Maine Et Loire
  - Centre de cancerologie les Dentellieres, Valenciennes, Nord
  - Centre Leon Berard, Lyon, Rhone
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - Institut Sainte Catherine, Avignon, Vaculuse
  - Hôpital d'Instruction des Armees Begin, Saint-Mandé, Val De Marne
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - Institut Curie - site de Paris, Paris
  - Hôpital Saint-Louis, Paris
  - Hopital Tenon, Paris
- Germany (7):
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Rotkreuzklinikum Muenchen gGmbH, Munich, Bavaria
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf, North Rhine-Westphalia
  - Haematologisch-Onkologische Schwerpunktpraxis, Troisdorf, North Rhine-Westphalia
  - Marienhospital Bottrop gGmbH, Bottrop, Rhineland-Palatinate
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck, Schleswig-Holstein
- Hong Kong (2):
  - The Chinese, Hong Kong
  - The University of Hong Kong, Shatin
- Italy (16):
  - Azienda Ospedaliera Universitaria Arcispedale Sant'Anna, Cona, Ferrara
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), U.O Oncologia Medica, Monza, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - IRCCS Centro di Riferimento Oncologico, Aviano, Pordenone
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Istituto Nazionale per la Ricerca sul Cancro di Genova, Genova
  - Azienda Ospealiera della Provincia di Lecco, Lecco
  - Azienda Ospedaliera Ospedali Riuniti Papardo-Piemonte, Messina
  - Ospedale San Raffaele, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - A.O.U. Policlinico di Modena, Modena
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Japan (17):
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-Ku, Tokyo-To
  - Aichi Cancer Center Hospital, Aichi
  - NHO Shikoku Cancer Center, Ehime
  - NHO Kyushu Cancer Center, Fukuoka
  - Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - NHO Hokkaido Cancer Center, Hokkaido
  - Kanagawa Cancer Center, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Niigata Cancer Center, Niigata
  - Okayama University Hospital, Okayama
  - NHO Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Saitama Cancer Center, Saitama
  - Shizuoka Cancer Center, Shizuoka
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Showa University Hospital, Tokyo
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (17):
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Virgen Macarena, Seville, Sevill
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - IOB-Institute of Oncology, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
- Taiwan (5):
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation, Sun Yat-Sen Cancer Center, Taipei
- United Kingdom (10):
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - Aberdeen Royal Infirmary, Aberdeen, Grampian Region
  - Queen Mary University of London, London, Greater London
  - University College London Hospitals, London, Greater London
  - Guy's Hospital, London, Greater London
  - Sarah Cannon Research Institute UK, London, Greater London
  - The Christie Hospital, Manchester, Greater Manchester
  - Western General Hospital, Edinburgh, Lothian Region
  - Nottingham University Hospitals City Campus, Nottingham, Nottinghamshire
  - Royal Surrey County Hospital, Guildford, Surrey

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Iwata H, Xu B, Kim SB, Chung WP, Park YH, Kim MH, Tseng LM, Chung CF, Huang CS, Kim JH, Chiu JWY, Yamashita T, Li W, Egorov A, Nishijima S, Nakatani S, Nishiyama Y, Sugihara M, Cortes J, Im SA. Trastuzumab deruxtecan versus trastuzumab emtansine in Asian patients with HER2-positive metastatic breast cancer. Cancer Sci. 2024 Sep;115(9):3079-3088. doi: 10.1111/cas.16234. Epub 2024 Jul 9. PMID 38979893
- [Derived] Cortes J, Hurvitz SA, Im SA, Iwata H, Curigliano G, Kim SB, Chiu JWY, Pedrini JL, Li W, Yonemori K, Bianchini G, Loi S, Borges GS, Wang X, Bachelot T, Nakatani S, Ashfaque S, Liang Z, Egorov A, Hamilton E. Trastuzumab deruxtecan versus trastuzumab emtansine in HER2-positive metastatic breast cancer: long-term survival analysis of the DESTINY-Breast03 trial. Nat Med. 2024 Aug;30(8):2208-2215. doi: 10.1038/s41591-024-03021-7. Epub 2024 Jun 2. PMID 38825627
- [Derived] Ma R, Shi Y, Yan R, Yin S, Bu H, Huang J. Efficacy and safety of trastuzumab deruxtecan in treating human epidermal growth factor receptor 2-low/positive advanced breast cancer:A meta-analysis of randomized controlled trials. Crit Rev Oncol Hematol. 2024 Apr;196:104305. doi: 10.1016/j.critrevonc.2024.104305. Epub 2024 Mar 3. PMID 38442809
- [Derived] Cortes J. Trastuzumab Deruxtecan versus Trastuzumab Emtansine for Breast Cancer: a plain language summary of the DESTINY-Breast03 study. Future Oncol. 2024 Feb;20(4):167-178. doi: 10.2217/fon-2023-0422. Epub 2023 Dec 7. PMID 38059424
- [Derived] Rugo HS, Crossno CL, Gesthalter YB, Kelley K, Moore HB, Rimawi MF, Westbrook KE, Buys SS. Real-World Perspectives and Practices for Pneumonitis/Interstitial Lung Disease Associated With Trastuzumab Deruxtecan Use in Human Epidermal Growth Factor Receptor 2-Expressing Metastatic Breast Cancer. JCO Oncol Pract. 2023 Aug;19(8):539-546. doi: 10.1200/OP.22.00480. Epub 2023 May 19. PMID 37207306
- [Derived] Curigliano G, Dunton K, Rosenlund M, Janek M, Cathcart J, Liu Y, Fasching PA, Iwata H. Patient-reported outcomes and hospitalization data in patients with HER2-positive metastatic breast cancer receiving trastuzumab deruxtecan or trastuzumab emtansine in the phase III DESTINY-Breast03 study. Ann Oncol. 2023 Jul;34(7):569-577. doi: 10.1016/j.annonc.2023.04.516. Epub 2023 May 12. PMID 37179020
- [Derived] Hurvitz SA, Hegg R, Chung WP, Im SA, Jacot W, Ganju V, Chiu JWY, Xu B, Hamilton E, Madhusudan S, Iwata H, Altintas S, Henning JW, Curigliano G, Perez-Garcia JM, Kim SB, Petry V, Huang CS, Li W, Frenel JS, Antolin S, Yeo W, Bianchini G, Loi S, Tsurutani J, Egorov A, Liu Y, Cathcart J, Ashfaque S, Cortes J. Trastuzumab deruxtecan versus trastuzumab emtansine in patients with HER2-positive metastatic breast cancer: updated results from DESTINY-Breast03, a randomised, open-label, phase 3 trial. Lancet. 2023 Jan 14;401(10371):105-117. doi: 10.1016/S0140-6736(22)02420-5. Epub 2022 Dec 7. PMID 36495879
- [Derived] Rugo HS, Bianchini G, Cortes J, Henning JW, Untch M. Optimizing treatment management of trastuzumab deruxtecan in clinical practice of breast cancer. ESMO Open. 2022 Aug;7(4):100553. doi: 10.1016/j.esmoop.2022.100553. Epub 2022 Aug 11. PMID 35964548
- [Derived] Cortes J, Kim SB, Chung WP, Im SA, Park YH, Hegg R, Kim MH, Tseng LM, Petry V, Chung CF, Iwata H, Hamilton E, Curigliano G, Xu B, Huang CS, Kim JH, Chiu JWY, Pedrini JL, Lee C, Liu Y, Cathcart J, Bako E, Verma S, Hurvitz SA; DESTINY-Breast03 Trial Investigators. Trastuzumab Deruxtecan versus Trastuzumab Emtansine for Breast Cancer. N Engl J Med. 2022 Mar 24;386(12):1143-1154. doi: 10.1056/NEJMoa2115022. PMID 35320644

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 524 participants were enrolled and treated at study sites in 14 countries. Primary results reported is from first participant randomized up to data cut-off date of 21 May 2021. The results presented are based on primary analysis up to 33 months. Data collection is still on-going and additional results will be provided after study completion.
Period: Overall Study
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Ado-trastuzumab Emtansine (T-DM1)
Started | 261 | 263
Completed | 136 | 49
Not Completed | 125 | 214
Not completed — Progressive Disease | 66 | 158
Not completed — Clinical Progression | 4 | 12
Not completed — Adverse Event | 35 | 17
Not completed — Withdrawal by Subject (from treatment only) | 13 | 11
Not completed — Lack of Efficacy | 3 | 3
Not completed — Physician Decision | 2 | 8
Not completed — Miscellaneous | 2 | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Full Analysis Set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Ado-trastuzumab Emtansine (T-DM1) | Total
Number analyzed (Participants) | 261 | 263 | 524
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 212 | 206 | 418
  >=65 years | 49 | 57 | 106
Age, Continuous [Median (Standard Deviation); unit: years] | 54.5 (11.11) | 54.2 (11.84) | 54.4 (11.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 260 | 262 | 522
  Male | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 152 | 162 | 314
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 9 | 19
  White | 71 | 72 | 143
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 26 | 20 | 46

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Based on Blinded Independent Central Review (BICR) in Participants With HER2-Positive, Unresectable and/or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane
Description: Progression-free survival (PFS) by BICR was defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Up to 33 months (data cut-off)
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set at data cut-off date of 21 May 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Ado-trastuzumab Emtansine (T-DM1)
Number analyzed (Participants) | 261 | 263
months | NA [18.5 to NA] — Median and upper CI was not estimable due to insufficient number of events. | 6.8 [5.6 to 8.2]

2. Secondary Outcome: Overall Survival (OS) in Participants With HER2-Positive, Unresectable and/or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane
Description: Overall survival (OS) was defined as the time from the date of first dose of study drug to the date of death due to any cause.
Time Frame: Up to 33 months (data cut-off)
Population: Overall survival (OS) was assessed in the Full Analysis Set at data cut-off date of 21 May 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Ado-trastuzumab Emtansine (T-DM1)
Number analyzed (Participants) | 261 | 263
months | NA [NA to NA] — Median and 95% CI was not estimable due insufficient number of events. | NA [NA to NA] — Median and 95% CI was not estimable due insufficient number of events.

3. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR) Based on BICR and Investigator Assessment in Participants With HER2-Positive, Unresectable and/or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane
Description: The Objective Response Rate (ORR) was defined as the percentage of participants who achieved a best overall response of confirmed Complete Response (CR) or Partial Response (PR), assessed by BICR and investigator assessment based on RECIST version 1.1. CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions. Confirmed ORR is reported.
Time Frame: Up to 33 months (data cut-off)
Population: Objective response rate was assessed in the Full Analysis Set at data cut-off date of 21 May 2021.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Ado-trastuzumab Emtansine (T-DM1)
Number analyzed (Participants) | 261 | 263
Percentage of Participants
  BICR | 79.7 [74.3 to 84.4] | 34.2 [28.5 to 40.3]
  Investigator Assessment | 77.0 [71.2 to 82.0] | 36.9 [31.0 to 43.0]

4. Secondary Outcome: Duration of Response (DoR) Based on BICR and Investigator Assessment in Participants With HER2-Positive, Unresectable and/or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane
Description: Duration of Response (DoR) was defined as the time from the date of the first documentation of objective response (complete response [CR] or partial response [PR]) to the date of the first objective documentation of progressive disease (PD) or death due to any cause. DoR in participants with confirmed CR/PR based on BICR and investigator assessment is reported.
Time Frame: Up to 33 months (data cut-off)
Population: Duration of Response (DoR) was assessed in the Full Analysis Set of participants with confirmed CR/PR at data cut-off date of 21 May 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Ado-trastuzumab Emtansine (T-DM1)
Number analyzed (Participants) | 261 | 263
months
  BICR: number analyzed (Participants) | 208 | 90
  BICR | NA [20.3 to NA] — Median and upper CI was not estimable due insufficient number of events. | NA [12.6 to NA] — Median and upper CI was not estimable due insufficient number of events.
  Investigator Assessment: number analyzed (Participants) | 201 | 97
  Investigator Assessment | NA [20.8 to NA] — Median and upper CI was not estimable due insufficient number of events. | NA [14.1 to NA] — Median and upper CI was not estimable due insufficient number of events.

5. Secondary Outcome: Progression-Free Survival (PFS) Based on Investigator Assessment in Participants With HER2-Positive, Unresectable and/or Metastatic Breast Cancer Previously Treated With Trastuzumab and Taxane
Description: Progression-free survival (PFS) by investigator assessment was defined as the time from the date of enrollment to the earlier of the dates of the first objective documentation of disease progression (as per RECIST v1.1) or death due to any cause. Progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions.
Time Frame: Up to 33 months (data cut-off)
Population: Progression-free survival (PFS) was assessed in the Full Analysis Set at data cut-off date of 21 May 2021.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Ado-trastuzumab Emtansine (T-DM1)
Number analyzed (Participants) | 261 | 263
months | 25.1 [22.1 to NA] — Upper CI was not estimable due to insufficient number of events. | 7.2 [6.8 to 8.3]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of signing the informed consent form up to 47 days after last dose of the study drug, up 33 months.
Description: A Treatment-emergent adverse event (TEAE) is defined as an AE that occurs, having been absent before the first dose of study drug, or has worsened in severity or seriousness after the initiating the study drug until 47 days after last dose of the study drug.
Arm/Group | Trastuzumab Deruxtecan (T-DXd) | Ado-trastuzumab Emtansine (T-DM1)
All-Cause Mortality (participants affected / at risk) | 33/257 | 53/261
Serious Adverse Events (participants affected / at risk) | 49/257 | 47/261
Other Adverse Events (participants affected / at risk) | 256/257 | 249/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Deruxtecan (T-DXd) (N=257) | Ado-trastuzumab Emtansine (T-DM1) (N=261)
Vomiting (Gastrointestinal disorders) | 5 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pneumonia (Infections and infestations) | 4 | 5
Pyrexia (General disorders) | 4 | 0
Disease progression (General disorders) | 3 | 1
Urinary tract infection (Infections and infestations) | 3 | 1
Anaemia (Blood and lymphatic system disorders) | 2 | 3
Cellulitis (Infections and infestations) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Seizure (Pregnancy, puerperium and perinatal conditions) | 2 | 0
COVID-19 (Infections and infestations) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pneumonitis (Infections and infestations) | 1 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Rhegmatogenous retinal detachment (Eye disorders) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Sudden death (General disorders) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Vasogenic cerebral oedema (Nervous system disorders) | 1 | 0
Platelet count decreased (Investigations) | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Angiodysplasia (Vascular disorders) | 0 | 1
Arterial haemorrhage (Vascular disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Biopsy lymph gland (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Brain herniation (Injury, poisoning and procedural complications) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Fatigue (General disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hepatic atrophy (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hypercalcaemia of malignancy (Endocrine disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Otolithiasis (Ear and labyrinth disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trastuzumab Deruxtecan (T-DXd) (N=257) | Ado-trastuzumab Emtansine (T-DM1) (N=261)
Nausea (Gastrointestinal disorders) | 195 | 79
Vomiting (Gastrointestinal disorders) | 126 | 26
Alopecia (Skin and subcutaneous tissue disorders) | 95 | 8
Constipation (Gastrointestinal disorders) | 88 | 51
Anaemia (Blood and lymphatic system disorders) | 83 | 43
Decreased appetite (Metabolism and nutrition disorders) | 75 | 44
Neutrophil count decreased (Investigations) | 75 | 25
Diarrhoea (Gastrointestinal disorders) | 75 | 18
Fatigue (General disorders) | 74 | 52
Aspartate aminotransferase increased (Investigations) | 66 | 105
White blood cell count decreased (Investigations) | 58 | 14
Alanine aminotransferase increased (Investigations) | 56 | 77
Platelet count decreased (Investigations) | 54 | 112
Headache (Nervous system disorders) | 54 | 38
Weight decreased (Metabolism and nutrition disorders) | 43 | 16
Neutropenia (Blood and lymphatic system disorders) | 41 | 7
Stomatitis (Infections and infestations) | 40 | 10
Blood alkaline phosphatase increased (Investigations) | 35 | 30
Hypokalaemia (Metabolism and nutrition disorders) | 33 | 26
Asthenia (General disorders) | 32 | 31
Dizziness (Nervous system disorders) | 32 | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29 | 42
Dyspepsia (Gastrointestinal disorders) | 29 | 16
Malaise (General disorders) | 29 | 10
Abdominal pain (Gastrointestinal disorders) | 29 | 5
Abdominal pain upper (Gastrointestinal disorders) | 28 | 12
Pyrexia (General disorders) | 27 | 39
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 26
Back Pain (Musculoskeletal and connective tissue disorders) | 24 | 16
Myalgia (Musculoskeletal and connective tissue disorders) | 23 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 23
Leukopenia (Blood and lymphatic system disorders) | 22 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 13
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 20 | 15
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 | 12
Peripheral sensory neuropathy (Nervous system disorders) | 19 | 25
Urinary tract infection (Infections and infestations) | 19 | 13
Pneumonia (Infections and infestations) | 18 | 9
Anxiety (Psychiatric disorders) | 18 | 6
Pneumonitis (Infections and infestations) | 18 | 1
Blood lactate dehydrogenase increased (Investigations) | 17 | 35
Blood bilirubin increased (Investigations) | 17 | 13
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 | 12
Oedema peripheral (General disorders) | 17 | 9
Rash (Skin and subcutaneous tissue disorders) | 16 | 24
Insomnia (Psychiatric disorders) | 15 | 24
Dysgeusia (Nervous system disorders) | 15 | 8
Lymphopenia (Blood and lymphatic system disorders) | 15 | 6
Hypertension (Vascular disorders) | 14 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 4
Lymphocyte count decreased (Investigations) | 14 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 31
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 13 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT03529110/Prot_SAP_001.pdf